CLINICAL TRIAL: NCT06581120
Title: Assessment of Gastric Contents in Patients Taking Glucagon-Like Peptide-1 Receptor Agonists: a Prospective Observational Cross-sectional Study
Brief Title: GLP_1 RA Ultrasound Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0304
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Glucagon Like Peptide-1 (GLP-1; Delayed Gastric Emptying; Risk of Aspiration; Diabetes; Morbid Obesity
Keywords: GLP-1; Glucagon like Peptide 1; Aspiration; Gastric empty
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus; Obesity, Morbid | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GLP-1: Individuals currently taking glucagon like peptide receptors who have a surgery scheduled with Cincinnati Children's Hospital same day surgery endocrinology clinic and will receive a point of care gastric ultrasound.
  Interventions: Drug: Glucagon-Like Peptide-1 receptor agonists; Diagnostic Test: Point of Care Gastric Ultrasound
- Control: Individuals not taking GLP-1 who have a surgery scheduled with Cincinnati Children's Hospital same day surgery or endocrinology clinic and will receive a point of care gastric ultrasound.
  Interventions: Diagnostic Test: Point of Care Gastric Ultrasound

INTERVENTIONS:
Drug: Glucagon-Like Peptide-1 receptor agonists — GLP-1 RAs: Glucagon like peptide-1 receptor agonists, this includes patients who are on Liraglutide, Semaglutide, Dulaglutide and Tirzepatide.Tirzepatide which is a combined GLP-1 RA/glucose-dependent insulinotropic polypeptide (GIP) agonist is included as a part of GLP-1 RAs.
  Groups: GLP-1
Diagnostic Test: Point of Care Gastric Ultrasound — A gastric ultrasound following a standard NPO period to determine gastric contents and risk of aspiration during surgery.
  Other Names: POGUS

SUMMARY:
The purpose of the study is to determine whether patients taking GLP-1 RAs have increased residual (left behind), gastric (stomach), contents due to delayed gastric emptying when following standard preoperative fasting guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index over 35
* Type 2 Diabetes
* Currently taking GLP01 RA agonist (for GLP 1 group)
* Not taking GLP-1 RA agonist (for control group)

Exclusion Criteria:

* Diagnosis of gastroparesis
* patient refusal to participate
* Previous gastric bypass or any other gastric surgery
* Currently on peritoneal dialysis
* Abdominal pathology
* Gastro-intestinal obstruction
* Pregnancy

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the endocrine clinic and from the preoperative surgical schedule.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Aspiration Risk determined by POGUS | Two years
  Difference between control group and GLP-1 group. Measured by Gastric contents during Point of Care Gastric Ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No